CLINICAL TRIAL: NCT04593394
Title: Inducible Laryngeal Obstruction in Severe Asthma
Brief Title: Inducible Laryngeal Obstruction in Severe Asthma in Severe Asthma
Status: Completed | Type: Observational
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 108266
Record Dates: First submitted 2020-10-13; First posted 2020-10-20 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-05

CONDITIONS: Asthma Chronic; Vocal Cord Dysfunction
Keywords: Inducible laryngeal dysfunction, Severe asthma,
MeSH Terms: conditions — Vocal Cord Dysfunction; Asthma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Severe asthma: Gina-guidlines treatment-step 5
  Interventions: Diagnostic Test: Continous laryngoscopy exercise test; Diagnostic Test: Overnight respiratory polygraphy
- Mild-moderate asthma: Gina-guidlines treatment-step 1-4
  Interventions: Diagnostic Test: Continous laryngoscopy exercise test; Diagnostic Test: Overnight respiratory polygraphy
- Subjects without asthma: Matches control-group without asthma
  Interventions: Diagnostic Test: Continous laryngoscopy exercise test; Diagnostic Test: Overnight respiratory polygraphy

INTERVENTIONS:
Diagnostic Test: Continous laryngoscopy exercise test — Participants walks on a tredmill with a a flexible naso-laryngoscope in the larynx allowing visulasion of the larynx and obstructions in the larynx at the epiglottic og glottic levels are scored
Diagnostic Test: Overnight respiratory polygraphy — Overnight respiratory polygraphy is a continuous recording of nasal airflow, thoracic and abdominal movements, heart rate and oxygen saturation during the night used to detected sleep apnoea

SUMMARY:
The first part will be a comparative cross-sectional study to identify the frequency of ILO and other comorbidites among participants with asthma compared to a group of reference subjects without asthma, matched for age- and gender and race.

The second part will be a longitudinally observational study study following participants for one year after the cross-sectional study. The Maat-scores ILO-symptoms and asthma-outcomes longitudinally will be evaluated, .

DETAILED DESCRIPTION:
Inducible laryngeal obstruction (ILO) is characterized by inappropriate closure of the structures of the larynx causing reduced airflow. The symptoms are breathing difficulties that resemble those seen in asthmatic patients, such as dyspnea, coughing and stridor. ILO may be diagnosed by the continuous laryngoscopy during exercise test (CLE-test), where the larynx is visualized live on video as the patient runs to exhaustion on a treadmill whilst having a laryngoscope placed through the nose.

The prevalence of ILO in asthmatic patients will be assesed by preforming a CLE-test twice in all participants at baseline and again after one year. Participant will be given visual feedback and instructed in breathing techniques. Others common comorbidities will be assessed by questionnaires and clinical interview. All patients with asthma will have a respiratory polygraph recording.

Changes in ILO-symptoms and asthma-symptoms and outcomes will be assessed after 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients with severe asthma (GINA 5)
* Patients with mild-moderate well-treated asthma (GINA step 1-4)
* Agroup of age- and gender matched control subjects without asthma also aged 18- 70.
* The patients must have had a stable disease the last one month before performing the CLE-test

Exclusion Criteria:

* No have underlying neurologic disease.
* No known cancer in the lung-head-neck
* No known vocal cord pathology.
* No history of life-threatening asthma required hospitalization.

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The sample size of the cohort with severe asthma will be: All patients with severe asthma followed in our clinic for severe asthma estimated to be around 80 participants, of them, we hope to recruit at least 40 to perform the CLE-test, and we plan to recruit 40 participants with mild asthma and 40 age- and gender matched control subjects without asthma
Sampling Method: Non-Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Prevalence of ILO in the participants | One year
  Continues during exercise(CLE)-test score at 2 or more at glottis or supraglottic level (Score range 0 minimum -3 maximum) 3 is full closure, 0 i open.
Changes in continues during exercise (CLE-)-test score | One year
  The absolute change from baseline CLE-score (Score range 0 minimum -3 maximum). 3 is full closure in larynx, 0 is open.

SECONDARY OUTCOMES:
The prevalence of OSA in asthma patients with ILO. | One year
  Prevalence of mild ( apnea-hypopnea index (AHI )5-15 ) moderat (AHI 15-30) and severe (AHI > 30 )OSA in participents with asthma and ILO
Changes in asthma-controll score (ACT) | One year
  Changes of 3 points of ACT-score are considered a clinical relevant change, score (score range minimum 5, maximum 25)
Number of asthma-exercabations | One year
  Annual asthma exacerbation rate and the precentage of patients with at least one asthma exacerbation. Asthma exacerbations are defined as worsening of asthma symptoms, and in participants on stable regimen with oral glucocorticoids, a doubling of the dose for 3 or more days or the use of systemic glucocorticoids for at least 3 days or beeing hospitalized.
Changes in mini-Asthma quality of life (m-AQLQ) | One year
  Changes of 0.5 at m-AQLQ are considered a clinical relevant change

CONTACTS AND LOCATIONS:
Overall Officials: Sverre Lehmann, PhD, Principal Investigator — Haukeland University Hospital
Locations (1):
- Haukeland University Hospital, Bergen, Norway

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Rogde AJ, Lehmann S, Halvorsen T, Clemm HH, Roksund OD, Hufthammer KO, Kvidaland HK, Vollsaeter M, Andersen TM. Prevalence and impact of exercise-induced laryngeal obstruction in asthma: a study protocol for a cross-sectional and longitudinal study. BMJ Open. 2023 Jun 16;13(6):e071159. doi: 10.1136/bmjopen-2022-071159. PMID 37328176